CLINICAL TRIAL: NCT03506646
Title: Dietary Nitrate Supplementation and Thermoregulation During Exercise
Brief Title: Dietary Nitrate Supplementation and Thermoregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0201-18-FB
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: 1:1 randomized, cross-over, double-blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice-Placebo (Experimental): Subjects will be tested on two different days, first day will be baseline and Beetroot juice and second day will be Placebo. Testing will take place forty-minutes after Beetroot juice/placebo intake. There will be a 2-week washout between testing days.
  Interventions: Dietary Supplement: Beet root juice
- Placebo-Beetroot juice (Experimental): Subjects will be tested on two different days, first day will be baseline and Placebo and second day will be Beetroot juice. Testing will take place forty-minutes after placebo/beetroot juice intake. There will be a 2-week washout between testing days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Placebo — Participants will be given a gelatin tablet to serve as the control condition. This will be a double-blinded, randomized, cross-over design to examine the effects of beetroot juice on endothelial function, leg function, and thermoregulation.
  Arms: Placebo-Beetroot juice
Dietary Supplement: Beet root juice — Beet root juice serves as a mode of dietary nitrate supplementation. This will be a double-blinded, randomized, cross-over design to examine the effects of beetroot juice on endothelial function, leg function, and thermoregulation.
  Arms: Beetroot juice-Placebo

SUMMARY:
This is a double-blinded, randomized, crossover design study to assess the effects of dietary nitrate supplementation (beetroot juice) on peripheral artery disease (PAD) patients (ages 50-85) diagnosed with Fontaine stage I or II PAD (as determined by vascular surgeon at UNMC). Exclusion criteria include: 1) experience severe claudication (leg pain) at rest or tissue loss due to PAD (Fontaine stage III and IV), 2) have limited walking capacity due to conditions other than PAD, 3) are already supplementing with a form of dietary nitrate, or 4) have an allergy to beetroot juice.

Subjects will be required to visit the lab 3 times and will be randomized to receive either the supplement or the placebo for the 2nd and 3rd visits. There will be a washout period of 14 days between the 2nd and 3rd visits. Visit 1 will take approximately 2 hours and the 2nd/3rd visits will take approximately 1.5 hours. Total experimentation period will last approximately 15 days.

Visit 1 will consist of non-invasive baseline testing including assessment of endothelial function (flow-mediated dilation by ultrasound imaging), maximal walking capacity (Gardner treadmill protocol), leg function (near-infrared spectroscopy, time to onset claudication, blood flow to lower extremities), and body core temperature (rectal thermometer). Visits 2 and 3 will require consumption of either the supplement or placebo. The same tests from the baseline measurements will be performed for visits 2 and 3. There will be a recommended fourth visit, albeit not required, to review study results.

DETAILED DESCRIPTION:
Background and rationale The vast majority of the research involving dietary nitrate supplementation, namely beetroot juice, has been performed mostly on samples of healthy populations. A few clinical populations have been studied, including heart failure with preserved ejection fraction, chronic obstructive pulmonary disease (COPD), and peripheral artery disease (PAD). In various populations, beetroot juice (BRJ) has been shown to decrease overall blood pressure, increase blood flow, increase muscle tissue oxygenation, improve body core temperature regulation, and increase exercise tolerance while decreasing the oxygen cost of exercise.

Blood pressure BRJ supplementation has been shown to have an immediate effect on reducing blood pressure, with the most substantial decreases recorded within approximately 2.5-3 hours following supplement consumption [1, 2]. Systolic, diastolic, and mean arterial blood pressures showed decreases of 10.4±3 mmHg, 8.1±2.1 mmHg, and 8.0±2.1 mmHg, respectively, in healthy volunteers [2]. During exercise in healthy individuals, systolic blood pressure remained lower throughout varying exercise intensities [1]. Blood pressure was also reduced in heart failure with preserved ejection fraction patients. After an acute dose of BRJ, resting systolic blood pressure significantly decreased when compared to placebo conditions (BRJ 127 ± 14 mmHg; placebo134 ± 14 mmHg) [3]. A slight reduction in systolic blood pressure during exercise may be beneficial to PAD patients. Hypertension, or high blood pressure, is a major risk factor for the development of PAD [4]. Decreasing overall blood pressure and slightly decreasing systolic blood pressure in response to light activity would result in a decrease in unnecessary stress placed on the cardiovascular system at rest and during exercise.

In a study involving PAD patients where 7 of the 8 participants were classified as either hypertensive or prehypertensive, BRJ consumption caused a significant reduction in diastolic blood pressure during rest that was maintained during exercise testing [5]. The study concludes that their data suggest that BRJ supplementation reduces blood pressure in PAD patients and this effect is maintained throughout exercise [5].

Oxygen delivery and muscle tissue oxygenation Oxygen demand of working muscle increases as activity level increases the efficiency of oxygen delivery and oxygen utilization is crucial to muscle function, as well as a necessary increase in blood flow. This is especially important in PAD patients; increasing oxygenation to areas of skeletal muscle ischemia may increase physical function. By using near-infrared spectroscopy, muscle tissue oxygenation can be examined. During cycling in healthy males supplementing with BRJ, the right vastus lateralis muscle oxyhemoglobin concentrations were greater than that of the placebo condition [6]. While cycling at a moderate intensity, the male cyclists had a 13% reduction in deoxyhemoglobin concentration amplitude post-supplementation, which indicated a reduction in fractional oxygen extraction in the right vastus lateralis muscle [6]. These results suggest that BRJ supplementation may promote a better balance between localized oxygen delivery and utilization as an index of muscle fractional oxygen extraction [6]. Overall, BRJ supplementation has been shown to increase working muscle tissue oxygenation during exercise.

In PAD patients, the oxygenation of the gastrocnemius with the worst PAD symptoms was monitored during a walking cardiopulmonary exercise test. Subjects showed a 48% reduction in deoxyhemoglobin concentration amplitude following BRJ supplementation, which indicated that fractional oxygen extraction was reduced [5]. During the exercise protocol, deoxyhemoglobin amplitude measures for the BRJ supplementation group at 100 and 200 seconds into exercise were reduced by 44% and 53%, respectively [5]. This response implies that BRJ supplementation in PAD patients improves a balance between local oxygen delivery and utilization as an index of muscle fractional oxygenation extraction by the working muscle. Increasing oxygenation to areas of skeletal muscle ischemia in PAD patients may increase physical function, but in order for this to be as efficient as possible, a dose-response relationship must be determined.

Blood flow and thermoregulatory response Increases in activity and oxygen demand of working skeletal muscle necessitate increases in blood flow. In PAD patients, increasing blood flow to working muscle becomes difficult due to atherosclerotic occlusions in the lower extremity arteries. Research in healthy populations showed significant increases in forearm blood flow during hand grip exercise in hypoxic conditions following an acute dosage of BRJ in comparison to placebo (BRJ 373 ± 38 mL/min; placebo 343 ± 32 mL/min).

Nitric oxide signals smooth muscle within the blood vessels (endothelium) to relax, which in turn increases blood flow to the localized area of vasodilation. In healthy populations, dietary nitrate supplementation increases vasodilation near the surface of the skin [7]. This increase in vasodilatory capacity and blood flow would create a stronger temperature gradient at the level of the skin, which would facilitate more efficient heat exchange as blood is cooled at the level of the skin (sweat evaporative, conductive, and convective cooling), causing decreased strain on the body.

In PAD patients, nitrite-related nitric oxide signaling showed to increase peripheral blood flow to hypoxic tissue, which is supported by a decrease in gastrocnemius deoxygenation and a decrease in blood pressure [5]. However, during brachial artery flow mediated dilation, peak dilation did not significantly change (BRJ 42.6 ± 10.6 seconds; placebo 41.0 ± 10.39 seconds), which suggested that endothelial production of nitric oxide did not change [5]. The unchanging vasodilatory response is likely due to the study not examining a BRJ dose-response relationship and its effects on vasodilation.

Exercise tolerance and oxygen cost BRJ supplementation has been shown to decrease oxygen cost during low-intensity and moderate-intensity exercise. In trained populations supplementing with BRJ, significant decreases in oxygen cost during the beginning stages of exercise have been detected [8, 9]. Oxygen cost during walking was shown to decrease by approximately 12% following BRJ supplementation [8]. BRJ supplementation showed a 20% decrease in oxygen cost during moderate-intensity cycling in recreationally trained men [10]. This reduction in oxygen cost implies an increase in exercise efficiency in light-to-moderate level exercise, which in turn increases exercise tolerance. In high-intensity exercise, time-to-exercise-failure increased by 15% following BRJ supplementation, which is also suggestive of an increase in exercise tolerance [8].

BRJ supplementation in clinical populations has also shown to improve exercise tolerance. In heart failure with preserved ejection fraction patients, submaximal endurance exercise improved by 24% following BRJ supplementation in comparison to placebo conditions (BRJ 449 ± 180 seconds; placebo 363 ± 125 seconds) [3]. In patients with COPD, walking distance increased by 11% and time to exercise fatigue increased by 6% [11]. In PAD patients, BRJ supplementation showed an 18% (32 second) increase to onset claudication pain and a 17% (65 seconds) increase peak walking time in comparison to placebo conditions [5]. These results in PAD patients show a substantial acute response to BRJ supplementation (~2 hours of consumption) during exercise testing.

In various populations, BRJ supplementation has shown to decrease blood pressure, improve blood flow, increase muscle tissue oxygenation, safely maintain core temperature, and increase exercise tolerance. The effects of BRJ specifically in PAD patients showed decreases in blood pressure, increases in time to onset claudication and exercise tolerance, but did not show a significant effect on endothelial function. Examining a dose-response relationship is necessary to determine the responses to BRJ supplementation (endothelial function, leg function, and blood vessel oxygen carrying capacity) in PAD patients.In this study, a higher dose of nitrate (280 mL, 16.8 mmol nitrates) will be examined [12]. BRJ supplementation has shown reductions in blood pressure, increased muscle tissue oxygenation, blood flow, and thermoregulatory response. These mechanisms all contribute to improving overall cardiovascular function. If these results are observed during this study, PAD patients may experience less claudication pain as well as better tolerance to daily physical activities and exercise.

ELIGIBILITY:
Inclusion Criteria:

1. be able to give written, informed consent
2. demonstrate positive history of chronic claudication
3. have a history of exercise-limiting claudication
4. have an ankle/brachial index < 0.90 at rest
5. have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks.
6. be between 50-85 years old

Exclusion Criteria:

1. pain at rest (severe claudication) and/or tissue loss due to PAD (Fontaine stage III and IV)
2. acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
3. limited walking capacity due to other conditions other than PAD
4. a form of nitrate supplementation already included in their diet/regimen
5. an allergy to beetroot juice

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liz Pekas, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vanhatalo A, Bailey SJ, Blackwell JR, DiMenna FJ, Pavey TG, Wilkerson DP, Benjamin N, Winyard PG, Jones AM. Acute and chronic effects of dietary nitrate supplementation on blood pressure and the physiological responses to moderate-intensity and incremental exercise. Am J Physiol Regul Integr Comp Physiol. 2010 Oct;299(4):R1121-31. doi: 10.1152/ajpregu.00206.2010. Epub 2010 Aug 11. PMID 20702806
- [Background] Webb AJ, Patel N, Loukogeorgakis S, Okorie M, Aboud Z, Misra S, Rashid R, Miall P, Deanfield J, Benjamin N, MacAllister R, Hobbs AJ, Ahluwalia A. Acute blood pressure lowering, vasoprotective, and antiplatelet properties of dietary nitrate via bioconversion to nitrite. Hypertension. 2008 Mar;51(3):784-90. doi: 10.1161/HYPERTENSIONAHA.107.103523. Epub 2008 Feb 4. PMID 18250365
- [Background] Eggebeen J, Kim-Shapiro DB, Haykowsky M, Morgan TM, Basu S, Brubaker P, Rejeski J, Kitzman DW. One Week of Daily Dosing With Beetroot Juice Improves Submaximal Endurance and Blood Pressure in Older Patients With Heart Failure and Preserved Ejection Fraction. JACC Heart Fail. 2016 Jun;4(6):428-37. doi: 10.1016/j.jchf.2015.12.013. Epub 2016 Feb 10. PMID 26874390
- [Background] Selvin E, Erlinger TP. Prevalence of and risk factors for peripheral arterial disease in the United States: results from the National Health and Nutrition Examination Survey, 1999-2000. Circulation. 2004 Aug 10;110(6):738-43. doi: 10.1161/01.CIR.0000137913.26087.F0. Epub 2004 Jul 19. PMID 15262830
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745
- [Background] Bailey SJ, Varnham RL, DiMenna FJ, Breese BC, Wylie LJ, Jones AM. Inorganic nitrate supplementation improves muscle oxygenation, O(2) uptake kinetics, and exercise tolerance at high but not low pedal rates. J Appl Physiol (1985). 2015 Jun 1;118(11):1396-405. doi: 10.1152/japplphysiol.01141.2014. Epub 2015 Apr 9. PMID 25858494
- [Background] Boegli Y, Gremion G, Golay S, Kubli S, Liaudet L, Leyvraz PF, Waeber B, Feihl F. Endurance training enhances vasodilation induced by nitric oxide in human skin. J Invest Dermatol. 2003 Nov;121(5):1197-204. doi: 10.1046/j.1523-1747.2003.12518.x. PMID 14708626
- [Background] Lansley KE, Winyard PG, Fulford J, Vanhatalo A, Bailey SJ, Blackwell JR, DiMenna FJ, Gilchrist M, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of walking and running: a placebo-controlled study. J Appl Physiol (1985). 2011 Mar;110(3):591-600. doi: 10.1152/japplphysiol.01070.2010. Epub 2010 Nov 11. PMID 21071588
- [Background] Larsen FJ, Weitzberg E, Lundberg JO, Ekblom B. Effects of dietary nitrate on oxygen cost during exercise. Acta Physiol (Oxf). 2007 Sep;191(1):59-66. doi: 10.1111/j.1748-1716.2007.01713.x. Epub 2007 Jul 17. PMID 17635415
- [Background] Bailey SJ, Winyard P, Vanhatalo A, Blackwell JR, Dimenna FJ, Wilkerson DP, Tarr J, Benjamin N, Jones AM. Dietary nitrate supplementation reduces the O2 cost of low-intensity exercise and enhances tolerance to high-intensity exercise in humans. J Appl Physiol (1985). 2009 Oct;107(4):1144-55. doi: 10.1152/japplphysiol.00722.2009. Epub 2009 Aug 6. PMID 19661447
- [Background] Leong P, Basham JE, Yong T, Chazan A, Finlay P, Barnes S, Bardin PG, Campbell D. A double blind randomized placebo control crossover trial on the effect of dietary nitrate supplementation on exercise tolerance in stable moderate chronic obstructive pulmonary disease. BMC Pulm Med. 2015 May 2;15:52. doi: 10.1186/s12890-015-0057-4. PMID 25934631
- [Background] Wylie LJ, Kelly J, Bailey SJ, Blackwell JR, Skiba PF, Winyard PG, Jeukendrup AE, Vanhatalo A, Jones AM. Beetroot juice and exercise: pharmacodynamic and dose-response relationships. J Appl Physiol (1985). 2013 Aug 1;115(3):325-36. doi: 10.1152/japplphysiol.00372.2013. Epub 2013 May 2. PMID 23640589

RESULTS

PARTICIPANT FLOW:
Groups:
- Beetroot Juice First, Then Placebo: Subjects will be tested on two different days. The first day will be beetroot juice and the second day will be a placebo. Testing will take place approximately one hour after intake. There will be a 14 day washout period between testing days.
  Beetroot juice: Beetroot juice serves as a mode of dietary nitrate supplementation. This will be a double-blinded, randomized, cross-over design to examine the effects of beetroot juice on endothelial function, leg function, and thermoregulation.
- Placebo First, Then Beetroot Juice: Subjects will be tested on two different days. The first day will be a placebo and the second day will be beetroot juice. Testing will take place approximately one hour after intake. There will be a 14 day washout period between testing days.
  Beetroot juice: Beetroot juice serves as a mode of dietary nitrate supplementation. This will be a double-blinded, randomized, cross-over design to examine the effects of beetroot juice on endothelial function, leg function, and thermoregulation.
Period: First Intervention (Day 1)
Arm/Group | Beetroot Juice First, Then Placebo | Placebo First, Then Beetroot Juice
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Beetroot Juice First, Then Placebo | Placebo First, Then Beetroot Juice
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Beetroot Juice First, Then Placebo | Placebo First, Then Beetroot Juice
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 11 patients with peripheral artery disease were recruited and assigned to the beetroot juice and placebo groups in a randomized crossover study design
Groups:
- Total: Total of all reporting groups
Arm/Group | Beetroot Juice First, Then Placebo | Placebo First, Then Beetroot Juice | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (7.26) | 70.80 (10.28) | 70.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Height [Mean (Standard Deviation); unit: cm] | 165.92 (16.10) | 160 (11.77) | 162.96 (13.94)
Weight [Mean (Standard Deviation); unit: kg] | 84.17 (17.34) | 68.54 (12.57) | 76.35 (14.95)
Hand grip strength [Mean (Standard Deviation); unit: kg] | 29.33 (14.75) | 29.60 (8.65) | 29.47 (11.70)
Body fat percentage [Mean (Standard Deviation); unit: % body fat] | 39 (10.22) | 35.7 (8.08) | 37.35 (9.15)
Resting Heart Rate [Mean (Standard Deviation); unit: beats per min] | 71.2 (8.9) | 68.2 (14.5) | 69.8 (11.2)
Resting Blood Pressure [Mean (Standard Deviation); unit: mm/Hg]
  Systolic blood pressure | 134 (11) | 127 (22) | 131 (16)
  Diastolic blood pressure | 82 (7) | 79 (5) | 80 (6)

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Endothelial Function
Description: Endothelial function will be assessed using flow mediated dilation to measure vasodilation in the brachial artery (baFMD).
Time Frame: Pre and post treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % dilation
Groups:
- Beetroot Juice: Participants will receive Beetroot juice supplementation.
- Placebo: Participants will receive the Placebo
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
% dilation
  Baseline | 4.34 (1.39) | 4.31 (1.26)
  Post Treatment | 5.6 (1.65) | 4.35 (1.24)

2. Secondary Outcome: Leg Endothelial Function
Description: Popliteal artery endothelial function will be measured using the flow mediated dilation (paFMD) technique to measure vasodilation with an ultrasound imaging system.
Time Frame: Pre and Post treatment
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: % dilation
Groups:
- Placebo: Participants will receive placebo.
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
% dilation
  Baseline | 2.45 (1.30) | 2.73 (1.46)
  Post Treatment | 4.11 (2.12) | 2.73 (1.46)

3. Secondary Outcome: Muscle Tissue Oxygenation
Description: Muscle tissue oxygenation will be assessed by using near-infrared spectroscopy (NIRS) during a maximal walking protocol. Assessment is measured in arbitrary units as mean changes in deoxygenated hemoglobin (HHb)
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: arbitrary units
Groups:
- Beetroot Juice: Participants will receive Beetroot juice.
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
arbitrary units
  Baseline | 7.19 (49.5) | 1.12 (30.1)
  Post Treatment | -9.48 (23.2) | 3.86 (26.7)

4. Secondary Outcome: Physical Walking Capacity
Description: Physical walking capacity will be measured during the Gardner treadmill protocol. Participants will walk on a treadmill at 2.0 mph. Grade will began at zero and will be increased by two percent every two minutes. Participants unable to walk at least 2.0 miles per hour (MPH) begin walking at 0.5 MPH and their speed is increased by 0.50 MPH every two minutes until the participant reaches 2.0 MPH. After reaching 2.0 MPH, treadmill grade is increased by two percent every two minutes. Participants are asked to continue walking without stopping until they cannot continue because of leg symptoms, exhaustion, or other symptoms.
Time Frame: maximum of 14 minutes each day for 2 days
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
meters
  Baseline | 368.3 (243.3) | 366.1 (245.6)
  Post treatment | 460.5 (279.3) | 361.8 (262.9)

5. Secondary Outcome: Autonomic Nervous System Activity
Description: Autonomic nervous system activity will be assessed using heart rate variability. Data represented as ratio between low frequency (LF) and high frequency (HF).
Time Frame: maximum of 60 minutes each day for 2 days
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
Ratio
  Baseline | 2.6 (0.8) | 2.4 (0.5)
  Post treatment | 2.1 (0.7) | 2.8 (0.6)

6. Secondary Outcome: Microvascular Function
Description: Microvascular function will be assessed using near-infrared spectroscopy. Changes in tissue oxygenation rate following reactive hyperemia will be denoted as % recovery rate used to interpret mitochondrial function.
Time Frame: maximum of 30 minutes each day for 2 days
Measure: Mean (Standard Deviation); unit: % recovery rate
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
% recovery rate
  Baseline | 24.74 (15.02) | 28.05 (17.95)
  Post treatment | 46.87 (18.18) | 30.13 (17.57)

7. Secondary Outcome: Blood Nitrate/Nitrite Levels
Description: Participants will have blood drawn from an antecubital vein using a vacutainer and needle (25 gauge) prior to baseline testing and experimental trial testing. This will be done to measure nitrate/nitrite levels at baseline, post beetroot juice (BRJ) intake, and post placebo intake.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: micromolar concentration
Arm/Group | Beetroot Juice | Placebo
Number analyzed (Participants) | 11 | 11
micromolar concentration
  Pre treatment | .22 (.09) | .27 (.16)
  Post Treatment | 1.54 (.44) | .25 (.17)

ADVERSE EVENTS:
Time Frame: 2 wk
Groups:
- Beetroot Juice: Subjects will be tested on two different days. The first day will be beetroot juice and the second day will be a placebo. Testing will take place approximately one hour after intake. There will be a 14 day washout period between testing days.
  Beetroot juice: Beetroot juice serves as a mode of dietary nitrate supplementation. This will be a double-blinded, randomized, cross-over design to examine the effects of beetroot juice on endothelial function, leg function, and thermoregulation.
- Placebo: Subjects will be tested on two different days. The first day will be a placebo and the second day will be beetroot juice. Testing will take place approximately one hour after intake. There will be a 14 day washout period between testing days.
  Beetroot juice: Beetroot juice serves as a mode of dietary nitrate supplementation. This will be a double-blinded, randomized, cross-over design to examine the effects of beetroot juice on endothelial function, leg function, and thermoregulation.
Arm/Group | Beetroot Juice | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT03506646/Prot_SAP_000.pdf